CLINICAL TRIAL: NCT01958268
Title: Dysphagia Handicap Index: A Structured Translation From English to German of a Quality of Life Questionnaire Relating to Swallowing
Brief Title: Dysphagia Handicap Index: A Structured Translation From English to German
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BJ_02_08_2013
Record Dates: First submitted 2013-09-19; First posted 2013-10-09 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pretest and validation of a translated questionnaire

SUMMARY:
Establishment of a questionnaire in German to determine in a structured and quantifiable manner the quality of life of patients with dysphagia.

ELIGIBILITY:
Inclusion criteria: All patients with dysphagia

Exclusion criteria: Inability to fill in the questionnaire

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from dysphagia
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients able to fully understand and fill out the german translation of the questionnaire. | Patients suffering from dysphagia for at least half a year will be asked to answer the questionnaire at the time of enrolment.
  Establishment of a questionnaire in german to determine in a structured and quantifiable manner the quality of life of patients with dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg E Bohlender, KD Dr. med., Principal Investigator — University Hospital Zurich, Division of Otorhinolaryngology
Locations (1):
- University Hospital Zurich, Division of Otorhinolaryngology, Zurich, Canton of Zurich, Switzerland